CLINICAL TRIAL: NCT02038426
Title: Ultrasonography Assessment of Peripheral Entheses in Axial Spondyloarthritis and in Healthy Subjects, Athletes or Not.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-A00759-36; 2013-27 (Other: AP HM)
Record Dates: First submitted 2013-08-01; First posted 2014-01-16 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Peripheral Entheses
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- the patients with SpA (Experimental)
  Interventions: Biological: BLOOD SAMPLES; Device: Radiographs of the sacroiliac joints; Device: Radiographs of heels; Device: SCAN
- sports subjects (Experimental)
  Interventions: Biological: BLOOD SAMPLES; Device: Radiographs of the sacroiliac joints; Device: Radiographs of heels; Device: SCAN
- control subjects (Other)
  Interventions: Biological: BLOOD SAMPLES; Device: Radiographs of the sacroiliac joints; Device: Radiographs of heels; Device: SCAN

INTERVENTIONS:
Biological: BLOOD SAMPLES
Device: Radiographs of the sacroiliac joints
Device: Radiographs of heels
Device: SCAN

SUMMARY:
Purpose:

* Assessment of ultrasound MASEI index in axial spondyloarthritis and in healthy subjects, athletes or not
* Comparison of the ultrasound semiology of enthesitis in the 3 populations
* Comparison of the MASEI scores in the 3 populations

ELIGIBILITY:
Inclusion Criteria:

* - Axial spondyloarthritis according to the ASAS classification criteria
* 18-45 years old
* Athletes are defined by sport activities greater than or equal to 6 hours per week
* Non athletes are defined by sport activities lesser than or equal to 1 hour per week

Exclusion Criteria:

* - History of heel or ankle surgery
* Recent corticosteroid infiltration of the heel or the ankle

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
enthesitis detection | 12 months
  Number of subject having at least an enthesitis in every group of subjects

SECONDARY OUTCOMES:
MASEI scores | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France